CLINICAL TRIAL: NCT00214526
Title: Multicenter Randomized Clinical Trial of the Alair System for the Bronchial Thermoplasty Treatment of Asthma
Brief Title: Asthma Intervention Research (AIR) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asthmatx, Inc. (Industry)
Responsible Party: Narinder S Shargill, PhD., Vice President, Clinical Affairs, Asthmatx, Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol #0602-20
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Results first posted 2010-10-18 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Asthma
Keywords: Asthma; Bronchial Thermoplasty; Airway Hyperresponsiveness
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alair Group (Experimental): Conventional therapy with ICS+LABA plus bronchial thermoplasty with the Alair System.
  Interventions: Procedure: Bronchial thermoplasty with the Alair System
- Control Group (Active Comparator): Conventional therapy with ICS+LABA.
  Interventions: Drug: Conventional therapy with ICS+LABA

INTERVENTIONS:
Procedure: Bronchial thermoplasty with the Alair System — Conventional therapy with ICS+LABA plus bronchial thermoplasty with the Alair System.
  Arms: Alair Group
Drug: Conventional therapy with ICS+LABA — Conventional therapy with ICS+LABA.
  Arms: Control Group

SUMMARY:
The purpose of this study is to demonstrate the effectiveness and safety of the Alair System for the treatment of asthma.

This will be a multicenter, randomized controlled study comparing the effects of treatment with the Alair System to standard drug therapy. One-hundred and ten subjects will be randomized 1:1 to either the Alair Group (Medical management + Alair treatment),or Control Group (Medical management only).

DETAILED DESCRIPTION:
Multicenter, randomized, controlled clinical trial conducted at 11 Investigational Sites in 4 countries (Canada, United Kingdom, Denmark, and Brazil).

Subjects underwent Baseline evaluations, Alair treatments or Control Visits, and follow-up evaluations at 12-Weeks, 6-Months, and 12-Months after the last Treatment or Control Visit. In order to maximize the power of the study, Baseline and Follow-up testing was conducted in 2 parts. In the first part subjects continued to take their asthma maintenance medications (inhaled corticosteroids (ICS) and long acting β2-agonists (LABA) during the test period. This is designated as the "ON-LABA" Phase. Following ON-LABA testing subjects were asked to abstain from LABA for the second part of the testing, and these results are designated as the "OFF-LABA" Phase.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adult; age 18-65 years
* Asthma requiring regular maintenance medication that includes inhaled corticosteroid (at least 200 μg beclomethasone per day or equivalent) AND long acting ß2 agonist (LABA) (at least 100 mg salmeterol per day or equivalent)
* Pre-bronchodilator FEV1 60-85% (patients stabilized on inhaled corticosteroids and long acting β2 agonists)
* PC20 < 8 mg/ml per methacholine inhalation test using standardized methods.
* Demonstration of worsening of asthma following 2-week withdrawal of LABA, as documented by either:
* an increase of at least 0.5 in the Juniper Asthma Control Questionnaire score, relative to the Questionnaire score in the 2 weeks preceding withdrawal of LABA, OR
* a decline of at least 5% in the average am Peak Expiratory Flow during the second week of LABA abstinence relative to the average am Peak Expiratory Flow during the week immediately preceding LABA withdrawal
* Non-smoker x 1 year or greater (if former smoker, less than 10 pack years total smoking history)
* Willingness and ability to give written Informed Consent
* Willingness and ability to comply with the study protocol, including requirements for taking and abstaining from medications.

Exclusion Criteria:

* Participation in another clinical trial involving respiratory intervention that could affect the outcome measures of this study, either within 6 weeks of the pretreatment evaluation, or during the study period
* Current or recent respiratory tract infection (resolved less than 6 weeks from pretreatment evaluation)
* History of recurrent (³ 3 infections/year) lower respiratory tract infection requiring antibiotics.
* With the exception of the use of a prophylactic bronchodilator for exercise, requirement for more than 4 puffs in a 24-hour period of a short-acting b2-adrenergic agonist such as albuterol or salbutamol 100 mg/puff or equivalent within the seven days immediately prior to commencement of Enrollment Testing, Part I.
* Unstable asthma as defined by the need for an extra visit to a healthcare provider, increase in or introduction of new maintenance or symptom relieving medications (including new requirement for IV or nebulized medications) within 6 weeks of enrollment
* Use of an internal or external pacemaker or internal cardiac defibrillator
* Significant co-morbid illness such as cancer, renal failure, liver disease or cerebral vascular disease
* POST-bronchodilator FEV1 of less than 65%.
* Known systemic hypersensitivity or contraindication to methacholine chloride or other parasympathomimetic agents
* Known sensitivity to medications required to perform bronchoscopy, including lidocaine, atropine and benzodiazepines
* Use of a systemic b-adrenergic blocking agent
* Pregnancy
* Nursing mother
* History of epilepsy
* Cardiovascular disease, including bradycardia, angina, cardiac dysrhythmia, conduction defect or cardiac myopathy
* Myocardial infarction or stroke within 6 months of the pretreatment evaluation
* Any active disease left untreated,
* Bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 125,000/mm2 or known coagulopathy (INR > 1.5)
* Use of anticoagulants
* Insulin-dependent diabetes
* Psychiatric disorder which in the judgement of the investigator could interfere with provision of informed consent, completion of tests, therapy, or follow-up
* Presence of segmental atelectasis, lobar consolidation, significant or unstable pulmonary infiltrate, or pneumothorax, confirmed on x-ray
* Interstitial lung disease
* Uncontrolled hypertension (>200 mmHg systolic or >100mmHg diastolic pressure)
* Known aortic aneurysm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2002-11; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narinder S Shargill, PhD, Study Director — Asthmatx, Inc.

REFERENCES:
- [Derived] Cox G, Thomson NC, Rubin AS, Niven RM, Corris PA, Siersted HC, Olivenstein R, Pavord ID, McCormack D, Chaudhuri R, Miller JD, Laviolette M; AIR Trial Study Group. Asthma control during the year after bronchial thermoplasty. N Engl J Med. 2007 Mar 29;356(13):1327-37. doi: 10.1056/NEJMoa064707. PMID 17392302

RESULTS

PARTICIPANT FLOW:
Groups:
- Alair Group: Conventional therapy with inhaled corticosteroids and long-acting beta-agonists (ICS+LABA) plus bronchial thermoplasty with the Alair System. Throughout the Treatment Period subjects maintained their baseline daily asthma maintenance medications regimen.
- Control Group: Conventional therapy with inhaled corticosteroids and long-acting beta-agonists (ICS+LABA). Throughout the Treatment Period subjects maintained their baseline daily asthma maintenance medications regimen.
Period: Randomized
Arm/Group | Alair Group | Control Group
Started | 56 | 56
Completed | 55 | 54
Not Completed | 1 | 2
Period: Treatment Period
Arm/Group | Alair Group | Control Group
Started | 55 | 54
Completed | 53 | 49
Not Completed | 2 | 5
Period: Post-Treatment Period
Arm/Group | Alair Group | Control Group
Started | 53 | 49
Completed | 52 | 49
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alair Group | Control Group | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.36 (11.18) | 41.65 (11.35) | 40.50 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 24 | 23 | 47
Region of Enrollment [Number; unit: participants]
  Canada | 21 | 21 | 42
  United Kingdom | 19 | 17 | 36
  Denmark | 3 | 4 | 7
  Brazil | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Mild Exacerbation Rate (OFF-LABA) (Change From Baseline)
Description: Average change from Baseline across 12-Week, 6-Month, and 12-Month (OFF-LABA) Follow-up visits. A mild exacerbation was defined as 2 consecutive days when at least one of the following occurs: 1. Morning peak expiratory flow falls at least 20% below the average morning peak flow recorded during the 7 days immediately prior to Enrollment testing; 2. More than 3 more puffs of rescue short acting bronchodilator are required than the average usage during the 7 days immediately prior to Enrollment testing; 3. Awakening at night with asthma symptoms.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Exacerbations/Subject/Week
Arm/Group | Alair Group | Control Group
Number analyzed (Participants) | 55 | 54
Exacerbations/Subject/Week | -0.16 (0.37) | 0.04 (0.29)

2. Secondary Outcome: Pre-Bronchodilator FEV1 (Percent Predicted) (Change From Baseline)
Description: Percent change from Baseline at 12-Weeks (ON-LABA) and 12-Weeks, 6-Months, and 12-Months (OFF-LABA) Follow-up Visits in pre-bronchodilator forced expiratory volume in 1 second (FEV1) (percent predicted).
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alair Group | Control Group
Number analyzed (Participants) | 55 | 54
Percent Change
  ON-LABA at 12 Weeks | 3.65 (17.54) | 0.32 (12.37)
  OFF-LABA at 12 Weeks | 5.28 (12.00) | 4.00 (24.22)
  OFF-LABA at 6 Months | 7.29 (15.58) | 5.17 (17.67)
  OFF-LABA at 12 Months | 8.33 (20.73) | 3.94 (20.49)

3. Secondary Outcome: Post-Bronchodilator FEV1 (Percent Predicted) (Change From Baseline)
Description: Percent change from Baseline at 12-Weeks (ON-LABA) and 12-Weeks, 6-Months, and 12-Months (OFF-LABA) Follow-up Visits in post-bronchodilator forced expiratory volume in 1 second (FEV1) (percent predicted).
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alair Group | Control Group
Number analyzed (Participants) | 55 | 54
Percent Change
  ON-LABA at 12 Weeks | -0.13 (12.03) | -0.13 (8.63)
  OFF-LABA at 12 Weeks | 0.76 (12.65) | 0.80 (16.01)
  OFF-LABA at 6 Months | 0.82 (11.67) | 0.13 (11.55)
  OFF-LABA at 12 Months | 0.89 (13.91) | 1.33 (13.08)

4. Secondary Outcome: Methacholine PC20 (Change From Baseline)
Description: Change from Baseline at 12-Weeks, 6-Months, and 12-Months (OFF-LABA) Follow-up Visits in "PC20" - provocative concentration of Provocholine (a brand of methacholine chloride) resulting in a drop of FEV1 of 20% or more from baseline. The patient inhales an aerosol of one or more concentrations of methacholine. The lower the concentration of methacholine that provokes a 20% (or greater) fall in FEV1, the more "responsive" or "hyperresponsive" the airways are. Conversely, a rise in methacholine PC20 indicates airways that have become less reactive.
Time Frame: Baseline, 12 Months
Measure: Geometric Mean (95% Confidence Interval); unit: mg/mL
Arm/Group | Alair Group | Control Group
Number analyzed (Participants) | 55 | 54
mg/mL
  OFF-LABA at 12 Weeks | 0.64 [0.37 to 1.09] | 0.37 [0.24 to 0.58]
  OFF-LABA at 6 Months | 0.50 [0.30 to 0.85] | 0.42 [0.25 to 0.70]
  OFF-LABA at 12 Months | 0.61 [0.36 to 1.03] | 0.50 [0.31 to 0.80]

5. Secondary Outcome: Peak Expiratory Flow (Morning and Evening) (Change From Baseline)
Description: Change from Baseline at 12-Weeks (ON-LABA) and 12-Weeks, 6-Months, and 12-Months (OFF-LABA) Follow-up Visits in morning and evening Peak Expiratory Flow (PEF). The peak expiratory flow rate measures the maximal rate at which a person can exhale air.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Alair Group | Control Group
Number analyzed (Participants) | 55 | 54
L/min
  Morning PEF: ON-LABA at 12 Weeks | 27.96 (48.98) | 1.37 (32.26)
  Morning PEF: OFF-LABA at 12 Weeks | 42.59 (41.77) | 12.98 (37.08)
  Morning PEF: OFF-LABA at 6 Months | 31.49 (42.48) | 7.39 (45.03)
  Morning PEF: OFF-LABA at 12 Months | 39.31 (48.74) | 8.52 (44.18)
  Evening PEF: ON-LABA at 12 Weeks | 29.85 (49.11) | 0.57 (32.51)
  Evening PEF: OFF-LABA at 12 Weeks | 38.23 (48.97) | 12.58 (32.69)
  Evening PEF: OFF-LABA at 6 Months | 29.38 (46.35) | 9.53 (41.39)
  Evening PEF: OFF-LABA at 12 Months | 37.70 (50.53) | 9.88 (40.95)

6. Secondary Outcome: Asthma Control Questionnaire (ACQ) Score (Change From Baseline)
Description: Change from Baseline at 12-Weeks (ON-LABA) and 12-Weeks, 6-Months, and 12-Months (OFF-LABA) Follow-up Visits in Asthma Control Questionnaire (ACQ) Score. The ACQ is a self-administered patient questionnaire that assesses individual subject asthma control. The ACQ comprises 6 questions that relate to the patient's asthma symptoms, activity limitations, and daily rescue bronchodilator use, and FEV1. Each question is scored from 0 (best) to 6 (worst) and averaged, resulting in a total score from 0 to 6. A decrease in the ACQ score indicates better asthma control.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alair Group | Control Group
Number analyzed (Participants) | 55 | 54
Units on a scale
  ON-LABA at 12 Weeks | -0.30 (0.77) | -0.01 (0.68)
  OFF-LABA at 12 Weeks | -1.15 (1.01) | -0.30 (1.02)
  OFF-LABA at 6 Months | -1.23 (0.98) | -0.51 (0.97)
  OFF-LABA at 12 Months | -1.18 (1.02) | -0.47 (1.00)

7. Secondary Outcome: Use of Rescue Medications (Change From Baseline)
Description: Change from Baseline at 12-Weeks (ON-LABA) and 12-Weeks, 6-Months, and 12-Months (OFF-LABA) Follow-up Visits in use of rescue medications (short acting bronchodilators) measured in puffs per week. Subjects recorded their use of rescue medication for asthma symptoms in their Daily Diary throughout the study.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Puffs/7 Days
Arm/Group | Alair Group | Control Group
Number analyzed (Participants) | 55 | 54
Puffs/7 Days
  ON-LABA at 12 Weeks | -3.62 (11.97) | 0.94 (12.10)
  OFF-LABA at 12 Weeks | -9.08 (15.59) | -2.56 (12.75)
  OFF-LABA at 6 Months | -5.84 (15.59) | -1.26 (14.10)
  OFF-LABA at 12 Months | -8.93 (17.21) | -1.17 (16.71)

8. Secondary Outcome: Use of Maintenance Medications (Change From Baseline)
Description: Change from Baseline at 12-Months (OFF-LABA) Follow-up Visit in use of maintenance medications (inhaled corticosteroids and/or long-acting beta-agonists).
Time Frame: Baseline, 12 Months
Measure: Number; unit: Subjects
Arm/Group | Alair Group | Control Group
Number analyzed (Participants) | 55 | 54
Subjects
  No Change in ICS Dosage | 52 | 52
  Increase in ICS Dosage | 1 | 1
  Decrease in ICS Dosage | 2 | 1

9. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ) Score (Change From Baseline)
Description: Change from Baseline at 12-Weeks (ON-LABA) and 12-Weeks, 6-Months, and 12-Months (OFF-LABA) Follow-up Visits in AQLQ score. The AQLQ consists of 32 questions (scale from 1 to 7, where 7 reflects a higher quality of life). The AQLQ score is the mean of the scores from the 32 individual questions. An increase in the AQLQ score indicates a better quality of life. A within-subject change in score of 0.5 represents the minimal important difference (MID).
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alair Group | Control Group
Number analyzed (Participants) | 55 | 54
Units on a scale
  ON-LABA at 12 Weeks | 0.48 (0.94) | 0.01 (0.90)
  OFF-LABA at 12 Weeks | 1.25 (1.18) | 0.29 (1.06)
  OFF-LABA at 6 Months | 1.23 (1.10) | 0.54 (1.06)
  OFF-LABA at 12 Months | 1.27 (1.01) | 0.58 (1.09)

10. Secondary Outcome: Total Symptom Score (Change From Baseline)
Description: Change from Baseline at 12-Weeks (ON-LABA) and 12-Weeks, 6-Months, and 12-Months (OFF-LABA) Follow-up Visits in Total Symptom Score. Total Symptom Score comprises the sum of six asthma symptom measurements. Each symptom is scored on a scale of 0 to 3 each day by the subject. The sum of the scores for these 6 symptoms comprises the Total Symptom Score, which measures overall asthma symptoms. The maximum score possible is 18. A lower Total Symptom score represents better asthma control.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alair Group | Control Group
Number analyzed (Participants) | 55 | 54
Units on a scale
  ON-LABA at 12 Weeks | -1.18 (2.16) | -0.33 (1.89)
  OFF-LABA at 12 Weeks | -1.73 (2.13) | -0.37 (2.24)
  OFF-LABA at 6 Months | -1.60 (2.13) | -0.66 (2.28)
  OFF-LABA at 12 Months | -1.91 (2.11) | -0.65 (2.48)

ADVERSE EVENTS:
Groups:
- Alair (Treatment Period): From first Treatment visit through 6 weeks after last Treatment visit.
- Control (Treatment Period): From first Control visit through 6 weeks after last Control visit.
- Alair (Post-Treatment Period): From 6 weeks after last Treatment visit through 1 year.
- Control (Post-Treatment Period): From 6 weeks after last Control visit through 1 year.
Arm/Group | Alair (Treatment Period) | Control (Treatment Period) | Alair (Post-Treatment Period) | Control (Post-Treatment Period)
Serious Adverse Events (participants affected / at risk) | 4/55 | 4/54 | 5/55 | 4/54
Other Adverse Events (participants affected / at risk) | 53/55 | 43/54 | 52/55 | 46/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alair (Treatment Period) (N=55) | Control (Treatment Period) (N=54) | Alair (Post-Treatment Period) (N=55) | Control (Post-Treatment Period) (N=54)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Collapse Of Lung (Partial Collapse Of Left Upper Lobe) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Lung Infection Pseudomonal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alair (Treatment Period) (N=55) | Control (Treatment Period) (N=54) | Alair (Post-Treatment Period) (N=55) | Control (Post-Treatment Period) (N=54)
Abnormal Chest Sound (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 4
Bronchial Irritation (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0
Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 16 | 10 | 11 | 7
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 14 | 3 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 10 | 21 | 19
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 3 | 2
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 | 17 | 26 | 28
Dyspnoea Exacerbated (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 3 | 3
Fatigue (General disorders) | 5 | 0 | 3 | 1
Headache (Nervous system disorders) | 15 | 10 | 15 | 14
Hypersensitivity (Immune system disorders) | 1 | 1 | 2 | 3
Influenza (Infections and infestations) | 0 | 1 | 3 | 1
Influenza Like Illness (General disorders) | 1 | 0 | 3 | 0
Migraine (Nervous system disorders) | 1 | 0 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 15 | 14
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 6 | 3
Nausea (Gastrointestinal disorders) | 8 | 3 | 5 | 0
Nocturnal Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 5 | 7 | 5
Oral Candidiasis (Infections and infestations) | 3 | 2 | 0 | 2
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 6 | 7
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 5 | 11 | 11
Pyrexia (General disorders) | 3 | 1 | 1 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5 | 2
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 5 | 9
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 2
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 9 | 1 | 4 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 3 | 0
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 10 | 3
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 34 | 7 | 16 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less